CLINICAL TRIAL: NCT04454411
Title: Brain Mechanisms of Cognitive Response to Pharmacotherapy in Opioid Use Disorder
Brief Title: Brain Mechanisms of Pharmacotherapy in Opioid Use Disorder
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Primary funding source has ended.
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 843403; NCT05596955 (obsolete NCT alias)
Record Dates: First submitted 2020-06-18; First posted 2020-07-01 (Actual); Results first posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2024-10

CONDITIONS: Opioid Dependence
Keywords: naltrexone; buprenorphine; neuroimaging
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine; vivitrol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Buprenorphine (Experimental): Participants assigned to treatment with extended-release buprenorphine
  Interventions: Drug: Brixadi
- Naltrexone (Active Comparator): Participants assigned to treatment with extended-release naltrexone
  Interventions: Drug: Vivitrol

INTERVENTIONS:
Drug: Brixadi — Extended release injectable Buprenorphine
  Other Names: Buprenorphine Injectable Product
  Arms: Buprenorphine
Drug: Vivitrol — Extended release injectable Naltrexone
  Other Names: Naltrexone Injectable Product
  Arms: Naltrexone

SUMMARY:
This study will investigate the mechanisms of cognitive-behavioral response to medications used for relapse prevention in opioid use disorder (opioid addiction, OUD), through investigation of the neural circuits underlying key cognition functions. The study will use previously validated cognitive probes, functional Magnetic Resonance Imaging (fMRI), and novel extended-release injectable preparations of opioid partial agonist buprenorphine and antagonist naltrexone, in OUD patients to explain the individual heterogeneity of OUD treatment response.

DETAILED DESCRIPTION:
This proposal seeks to identify the neural circuits underlying the cognitive effects of medication assisted therapy (MAT) for OUD. The study will examine the neurocognitive effects of MAT by comparing two preparations with different pharmacodynamic properties (extended release buprenorphine and naltrexone, XRBUP, XRNTX) in three key domains (incentive salience, executive functioning, and emotion processing) using task functional Magnetic Resonance Imaging (MRI). In the 1st phase of the study, forty treatment-seeking OUD patients will be randomized to XRNTX or XRBUP groups after detoxification. Participants will undergo medication induction followed by monthly injections and urine toxicology monitoring for 120 days. Neuroimaging will follow completion of detoxification (pre-treatment) and 15 days after the second injection (on-treatment). The second study phase will extend the paradigm to an independent sample of 160 additional participants and test the explanatory value of MAT-induced changes in the neuroimaging signal in the classification of OUD treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Males and Females
2. 18-65 Years old
3. OUD by DSM5 Criteria, confirmed by history and physical examination including urine toxicology, medical records and self-report
4. Opioids are the drug of choice
5. Interested in injectable extended release agonist or antagonist treatment
6. Have a stable address, working command of English language, and telephone access.
7. Women of childbearing age must use an effective contraceptive

Exclusion Criteria:

1. Psychiatric Co-morbidities:

   1. Lifetime diagnoses of any psychotic disorder, e.g. schizophrenia, schizoaffective disorder, bipolar disorder type 1.
   2. Psychiatric Co-morbidities: Psychiatric disorders requiring current medication treatment, e.g. moderate to severe depression. Mild to moderate Depressive and Anxiety disorders and Attention Deficit Hyperactivity Disorder that do not require prescription stimulants and DSM5 Cluster B and C personality disorders are also allowed.
   3. Polysubstance users whose drug of choice is not opioids.
2. Contraindications for XRNTX or XRBUP e.g. active liver disease.
3. Medical and surgical conditions such as malignancy that may affect patients' ability to receive XRNTX or XRBUP treatment because it may interfere with opioid analgesia
4. Contraindications for MRI, e.g. claustrophobia, indwelling foreign magnetic agents.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Loughead, Ph.D., Principal Investigator — University of Pennsylvania
Locations (1):
- 3535 Market Street, Suite 4100, University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 143 individuals contacted the study staff expressing interest in phone screening. Of these, 28 individuals completed phone screening and three were eligible for the study and consented. One of the consented individuals was later excluded due to risk of metal fragments in the body. Two participants were lost to follow-up prior to randomization.
Pre-assignment Details: One of the consented individuals was later excluded due to risk of metal fragments in the body. Two participants were lost to follow-up prior to randomization.
Period: Overall Study
Arm/Group | Buprenorphine | Naltrexone
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 143 individuals contacted the study staff expressing interest in phone screening. Of these, 28 individuals completed phone screening and three were eligible for the study and consented. One of the consented individuals was later excluded due to risk of metal fragments in the body. Two participants were lost to follow-up prior to randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | Buprenorphine | Naltrexone | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Continuous
Sex: Female, Male
Ethnicity (NIH/OMB)
Race (NIH/OMB)
COWS

OUTCOME MEASURES:

1. Primary Outcome: fMRI Signal
Description: Brain fMRI response to neurocognitive probes
Time Frame: up to 90 days
Population: as for baseline characteristics
Arm/Group | Buprenorphine | Naltrexone
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Urine Toxicology: Opioid
Description: Rapid semi-quantitative ELISA urine drug screen test for morphine, oxycodone and methadone, followed by (cut off levels):
  Methadone (MTD) Methadone 300 ng/mL Opiates (OPI 300) Morphine Morphine **300 ng/mL Oxycodone (OXY) Oxycodone 100 ng/mL
Time Frame: Through the study completion, up to 120 days
Population: as for baseline characteristics
Arm/Group | Buprenorphine | Naltrexone
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Anxiety
Description: Hamilton Anxiety Rating Scale (HAM-A) (Hamilton, 1967). The HAM-A is a 15-minute, 14-item, clinician-administered instrument that measures current anxiety and changes in anxiety symptoms. Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe.
Time Frame: Through the study completion, up to 120 days
Population: as for baseline characteristics
Arm/Group | Buprenorphine | Naltrexone
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Depression
Description: Hamilton Depression Rating Scale (HAM-D) (Hamilton, 1959 #2497). The HAM-D is a 20-minute, 24-item interview that measures the severity of depression and changes in depressive symptoms. HAM-D form includes 21 items, however the scoring is based on the first 17. Eight items are scored on a 5-point scale, ranging from 0 = not present to 4 = severe. Nine are scored from 0-2. The HAM-D score level corresponds to the clinical severity of depression as follows: 10 - 13 mild; 14-17 mild to moderate; >17 moderate to severe.
Time Frame: Through the study completion, up to 120 days
Population: as for baseline characteristics
Arm/Group | Buprenorphine | Naltrexone
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Non-opioid Urine Toxicology
Description: Rapid semi-quantitative ELISA urine drug screen test for amphetamine/methamphetamine, benzodiazepines, cocaine, phencyclidine, cannabinoids and cotinine, with cut off levels:
  Amphetamine/Methamphetamine 500/1000ng/ml Benzodiazepines Enzyme Immunoassay (EIA) 200 ng/mL Cocaine Metabolite (Benzoylecgonine) EIA 150/300 ng/mL Cotinine EIA 250 ng/mL Phencyclidine EIA 25 ng/mL THC (Cannabinoids) EIA 20/50 ng/mL*
Time Frame: Through the study completion, up to 120 days
Population: as for baseline characteristics
Arm/Group | Buprenorphine | Naltrexone
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Description: 143 individuals contacted the study staff expressing interest in phone screening. Of these, 28 individuals completed phone screening and three were eligible for the study and consented. One of the consented individuals was later excluded due to risk of metal fragments in the body. Two participants were lost to follow-up prior to randomization.
Arm/Group | Buprenorphine | Naltrexone
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-17): https://cdn.clinicaltrials.gov/large-docs/11/NCT04454411/Prot_SAP_000.pdf